CLINICAL TRIAL: NCT05869136
Title: Comparative Evaluation Of Microneedling Alone vs Microneedling Along With Hyaluronic Acid In Thin Gingival Phenotype: A Split Mouth Randomized Clinical Trial
Brief Title: Evaluation Of Microneedling Alone vs Microneedling Along With Hyaluronic Acid In Thin Gingival Phenotype
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Nishi Tanwar
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Thin-gingiva
MeSH Terms: interventions — Percutaneous Collagen Induction; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Microneedling along with hyaluronic acid in thin gingival phenotype
  Interventions: Procedure: microneedling and hyaluronic acid for increasing gingival thickness in thin gingival phenotype
- Control group (Active Comparator): Microneedling in thin gingival phenotype
  Interventions: Procedure: microneedling for increasing gingival thickness in thin gingival phenotype

INTERVENTIONS:
Procedure: microneedling and hyaluronic acid for increasing gingival thickness in thin gingival phenotype — All the participants will undergo phase-I therapy. Oral hygiene instructions will be imparted and will be reinforced at each appointment.
  Local anaesthesia in the form of xylocaine spray will be administered.
  Hyaluronic acid:
  HA will be injected in the attached gingiva and MN will be carried out 1mm below the gingival margin on the keratinized gingiva of the tooth to be treated with thirty-gauge (0.255 mm) lancet needles in the test group.
  Arms: Test group
Procedure: microneedling for increasing gingival thickness in thin gingival phenotype — All the participants will undergo phase-I therapy. Oral hygiene instructions will be imparted and will be reinforced at each appointment.
  Local anaesthesia in the form of xylocaine spray will be administered and microneedling alone will be performed in control group
  Arms: Control group

SUMMARY:
The periodontal phenotype has been defined as the combination of gingival phenotype and buccal bone plate thickness (bone morphotype).Periodontal phenotype cannot be fully assessed but gingival phenotype can be evaluated through a standard and reproducible way.

Gingival recession is usually observed in the presence of trauma and inflammation in individuals with thin phenotypes, whereas pocket formation has been reported in individuals with thick phenotypes.

Various soft tissue augmentation procedures include: sub-epithelial connective tissue graft, free gingival graft, modified roll technique and use of acellular dermal matrix. The drawbacks of these techniques include second surgical site creation, post-operative discomfort, time consuming procedure, etc.

Recent studies have shown i-PRF, microneedeling and hyaluronic acid procedures to be effective in increasing gingival tissue thickness.

HA has been widely used in the dental field, specially periodontology, due to its bacteriostatic, fungistatic, anti-inflammatory, anti-edematous, osteoinductive, and pro-angiogenetic properties. HA's role in tissue regeneration and wound healing has gained huge interest in recent studies.

Microneedling (MN) is also known as "percutaneous collagen induction therapy." Microinjuries created by MN result in minimal superficial bleedings and create a wound-healing cascade from which various growth factors, such as platelet-derived growth factors, transforming growth factors, connective tissue growth factor and fibroblast growth factors, are released.Study has shown a statistically significant increase in gingival thickness when microneedling was performed along with i-PRF in comparison to standalone i-PRF.

Few human trials have been conducted using MN and Hyaluronic acids in literature for gingival augmentation in thin periodontal phenotype. Considering the effects of MN and hyaluronic acid on the biological potential, neoangiogenesis, neocollagenesis and wound, the present Randomized clinical trial is designed to evaluate the effects of MN alone and MN along with hyaluronic acid in thin gingival phenotype.

DETAILED DESCRIPTION:
Gingival phenotype refers to gingival thickness (GT) and keratinized tissue width (KTW).

Gingival phenotypes can be classified as scalloped and thin or flat and thick gingiva. Thin gingival phenotype are very friable and might be prone to recede in response to traumatic insults, such as plaque-related inflammation and traumatic toothbrushing .Studies have believed that HA accelerates the wound healing process, and promotes regeneration, as it maintains the viability of oral fibroblasts, increases their proliferative and migratory abilities, and enhances the expression of genes encoding type III collagen and transforming growth factor-β. Study has shown a statistically significant increase in gingival thickness when microneedling was performed along with i-PRF in comparison to standalone i-PRF.

Given these characteristics,this study will be conducted to comparative evaluation of microneedling alone and along with hyaluronic acid on thin gingival phenotype.

The present randomized controlled clinical trial will be conducted in the department of periodontics and oral implantology,Post Graduate Institute of Dental Sciences,Rohtak.Study design is of 24 months.

Total 20 patients will be recruited on the basis of inclusion and exclusion criteria with thin periodontal phenotypes who had consulted to the Department of Periodontology, Post Graduate Institute of Dental Sciences, Rohtak.

20 systematically healthy patients having thin gingival phenotypes will be included in this split-mouth randomized controlled trial. For each patient, each side of the anterior mandible will be randomly allocated to one of the two procedures (MN or MN with Hyaluronic acid)using chit system. In the MN group microneedling will be done 1 mm below the gingival margin with 30-gauze lancet needles. In the HA with MN group, the selected sites of the gingiva will injected with cross-linked HA using a 30-gauge microneedle followed by microneedling. This described procedure will be repeated in both groups three times with intervals of 10 days. The GT, KTW, and periodontal indices: gingival index (GI), bleeding on probing (BOP), and probing depth (PD) will be measured at baseline, 1 month, 6 months and 9 months.

ELIGIBILITY:
Inclusion Criteria:

• Thin gingival phenotype with gingival tissue thickness <1mm in mandibular anteriors

All the patients will be subjected to phase-I therapy and will be included after achieving healthy gingiva with Plaque index (Silness & Loe) <1, gingival index (Loe & Silness) <1 and showing adequate compliance and willing to participate in the study.

Exclusion Criteria:

* Patients having systemic diseases such as hypertension, diabetes, hyperthyroidism or on medications that influence the outcome of periodontal procedure
* Smokers, tobacco users
* Previous periodontal surgery
* No haematological disorders.
* Use of blood thinners
* Use of any drugs that might lead to gingival enlargement
* Stress, bruxism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Measurement of gingival thickness (GT) | 9 months
  To measure GT from the apical 1.5 mm of the gingival margin, a No:15 endodontic spreader with a 3-mm-diameter silicone disc will be placed in the centre and will be measured on Vernier caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nishi Tanwar, MDS, Principal Investigator — Post graduate institute of dental sciences,Rohtak,Haryana,India
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India